CLINICAL TRIAL: NCT06607068
Title: Assessment of Taurine Concentration in Older Women With/Without Obesity And With/Without Type 2 Diabetes Mellitus: a Cross-Sectional Study
Brief Title: Assessment of Taurine Concentration in Older Women With/Without Obesity And With/Without Type 2 Diabetes Mellitus
Status: Active, not recruiting | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Adelino Sanchez Ramos da Silva, PhD, University of Sao Paulo
Other Study IDs: 75476423.4.0000.5659; 2023/15008-9 (Other Grant/Funding Number: Fundação de Amparo à Pesquisa do Estado de São Paulo)
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Obesity and Type 2 Diabetes
Keywords: diabetes mellitus; obesity; aging; taurine; oxidative stress
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples will be collected in the morning, after 12 hours of fasting, by experienced nurses. 5 ml of blood will be collected for analysis of biochemical markers (after centrifugation and separation of plasma/serum, they will be stored in a freezer at -80°C for analysis).
  The evaluation of biochemical markers will involve the quantification of insulin sensitivity, glycemia, HbA1c, total cholesterol, insulin, triglycerides and HDL cholesterol. The kits Liquiform Total Cholesterol, HDL Cholesterol, Liquiform Triglycerides and Liquiform Glucose from Labtest diagnóstica® will be used, using an enzymatic system and absorbance spectrophotometer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- GIObDM - Older women with obesity and type 2 diabetes mellitus: Obesity will be assessed using the Body Mass Index (BMI), with older women being considered obese if they have a BMI above 30 km/m² (OPAS, 2002)
  Interventions: Other: None (Observational study)
- GIOb - Older women with obesity and without type 2 diabetes mellitus: Obesity will be assessed using the Body Mass Index (BMI), with elderly women being considered obese if they have a BMI above 30 km/m² (OPAS, 2002)
  Interventions: Other: None (Observational study)
- GIDM - Older women without obesity and with type 2 diabetes mellitus: The groups with DM2 will include elderly women who have already been medically diagnosed with DM2 , have been using a hypoglycemic/antidiabetic medication for at least 6 months and have fasting blood glucose ≥ 126mg/dL and/or HbA1c ≥ 6.5% in a blood test in the last 6 months.
  Interventions: Other: None (Observational study)
- GIEut - Eutrophic older women: For the group of eutrophic older women, they must have a BMI ≥ 23 and ≤ 28 kg/m² (OPAS, 2002). The medications used by all participants will be surveyed, as well as their dosages and daily consumption.
  Interventions: Other: None (Observational study)

INTERVENTIONS:
Other: None (Observational study) — None (Observational study)

SUMMARY:
Aging is a multifactorial process marked by several epigenetic and molecular changes, such as telomere shortening, DNA exposure to damage, mitochondrial dysfunction, accumulation of senescent cells, and oxidative stress. Such changes lead to the degeneration of cells and molecules, which affects tissues, organs, and systems over time, reducing the human body's ability to resist damage and favoring the development of chronic diseases such as Type 2 Diabetes Mellitus (T2DM). Taurine, a semi-essential amino acid, appears to be related to oxidative homeostasis, glucose control, and inflammation. Therefore, knowing the plasma concentrations of this amino acid in different populations is necessary to obtain a better understanding of the role of taurine in the pathophysiology of obesity and T2DM in older population, in addition to generating hypotheses regarding interventions capable of attenuating oxidative stress and inflammation, which are important hallmarks of aging.

DETAILED DESCRIPTION:
The aim of this study is to investigate whether health status (women with obesity, T2DM and no comorbidities) promotes changes in plasma taurine concentration and to correlate this concentration with biochemical markers (e.g. blood glucose, total cholesterol, insulin, glycated hemoglobin, triglycerides and HDL cholesterol). As well as to evaluate and compare the physical capacities of the different groups. Methods: Forty older women will participate in the cross-sectional study and will be allocated into four distinct groups, and will be classified as follows: older women with obesity and T2DM, older women with obesity and no T2DM, older women without obesity and with T2DM; eutrophic older women, with 10 older women in each group. The following will be performed: body composition assessment by total and regional body scanning using iDXA, anthropometry, tests to assess physical performance, peripheral blood collection for analysis of biochemical markers and the Physical Activity Level will be assessed using the Modified Baecke Questionnaire for Olders. For statistical analysis, One-way ANOVA will be used to verify the differences and compare the four groups. Expected results: It is expected that older women with obesity and T2DM will have lower plasma taurine concentration and also lower performance in physical tests, compared to the other groups.

ELIGIBILITY:
Inclusion Criteria:

Have not exercised regularly for at least 3 months;

Exclusion Criteria:

1. use of insulin;
2. consumption of multivitamin supplements or antioxidant vitamins;
3. consumption of mineral supplements such as Copper, Zinc and/or Manganese;
4. liver disease;
5. chronic kidney disease;
6. coronary disease;
7. thyroid disorders;
8. infectious diseases;
9. regular consumption of alcoholic beverages;
10. smoking;
11. the Mini Mental State Examination (MMSE) will be applied, which has a total score ranging from 0-30 points. For the elderly women to be included in the study, they must have a score greater than or equal to 13 points

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The sample will consist of 40 elderly women who will be allocated into four distinct groups with 10 elderly women in each group.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Plasma taurine concentration | 1 day at baseline
  Collected in EDTA tubes, were centrifuged and the plasma taurine concentration was evaluated using HPLC (high performance liquid chromatography).

SECONDARY OUTCOMES:
Lipid Profile | 1 day at baseline
  Serum levels of HDL, total cholesterol and triglycerides will be assayed (mg/dL)
Glycemic Profile | 1 day at baseline
  Serum levels of estimated average blood glucose (mg/dL)
Glycated hemoglobin | 1 day at baseline
  Serum levels glycated hemoglobin (%)
Macronutrients intake | 1 day at baseline
  The participants dietary intake will be assessed using a three-day dietary recall. The records must be completed by the participants on two weekdays and one weekend day. The professional Dietbox software will be used to calculate the caloric intake of macronutrients
Microminerals intake | 1 day at baseline
  The participants dietary intake will be assessed using a food registry of 3 days. The records must be completed by the participants on two weekdays and one weekend day. The professional Dietbox software will be used to calculate the caloric intake of microminerals
Level of consumption of ultra-processed foods | 1 day at baseline
  This study will evaluate the level of consumption of ultra-processed foods. The NOVA classification will be used for this purpose.
Upper limb strength endurance test: forearm flexion | 1 day at baseline
  Upper limb strength endurance test: forearm flexion for 30 seconds; To assess the strength endurance of the upper limbs, the forearm flexion test will be applied. The number of repetitions in 30 seconds will be counted.
Sit-to-Stand-Test | 1 day at baseline
  Sit-to-Stand-Test (30 seconds). This test will be used to quantify the lower limb strength of older women, and is recommended in the literature for this population. The number of repetitions in 30 seconds will be counted.
Lower limb muscle strength on an adjustable isokinetic dynamometer. | 1 day at baseline
  The angular velocities that will be used in the test will be 60º/s. A series of ten repetitions will be performed for the dominant limb for familiarization, followed by a 3-minute rest.
Body fat percentage (%) | 1 day at baseline
  Using the total body scan from the Dual-energy X-ray absorptiometry (DXA), body fat percentage will be assessed
Six-minute walk test | 1 day at baseline
  This test aims to assess aerobic capacity. The 6-minute walk test uses a 45.7 m total rectangular path: 18.28 m long by 4.57 m wide. The participant will be instructed to walk as fast as possible (without running) during the 6 minutes, as many times as they can in the rectangle. At the end of the time, the evaluator will record the total distance covered by the participant in meters.
Measurement of manual grip strength | 1 day at baseline
  The older woman&amp;amp;amp;amp;#39;s forearm should be positioned in half pronation, with the wrist in a neutral position. The hand should be positioned on the dynamometer, which will be held by the evaluator. Three attempts will be made with the dominant hand, with 3 seconds of grip and one-minute intervals between them. Of the three attempts, the one with the highest peak force (the largest measurement) will be recorded, in kilograms of force.

CONTACTS AND LOCATIONS:
Overall Officials: Adelino Sanchez Ramos da Silva, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Escola de Educação Física e Esporte de Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No